CLINICAL TRIAL: NCT04360590
Title: Pressure Support Ventilation (PSV) Versus Neurally Adjusted Ventilatory Assist (NAVA) in Difficult to Wean Pediatric ARDS Patients: a Physiologic Crossover Study
Brief Title: Pressure Support Ventilation Versus Neurally Adjusted Ventilatory Assist in Difficult to Wean Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SPINAZZOLA GIORGIA, Medical doctor, specialist in Anesthesia and Intensive Care Medicine, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: A693/CE2010
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Distress Respiratory Syndrome; Weaning Failure
Keywords: patient-ventilator interaction; pediatric acute respiratory distress syndrome; difficult weaning
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pressure support ventilation versus neurally adjusted ventilatory assist — All patients underwent three mechanical ventilation modes, lasting 1 hour each: pressure support mode, neurally adjusted ventilatory assist and again pressure support ventilation

SUMMARY:
This study assessed the effects of NAVA versus Pressure Support Ventilation (PSV) on patient-ventilator interaction in pediatric patients with difficult weaning from mechanical ventilation after moderate Pediatric Acute Respiratory Distress Syndrome (PARDS).

DETAILED DESCRIPTION:
12 pediatric patients, admitted in Pediatric Intensive Care Unit (PICU) with moderate PARDS and who failed up to 3 SBTs in less than 7 days, were enrolled in this study. These patients underwent three studies conditions, lasting 1 hour each: Pressure support ventilation 1, Neurally adjusted ventilatory assist and Pressure support ventilation 2.

During each trial were recorded the patient tracings of flow, airway pressure and electrical activity of diaphragm for the patient-ventilator interaction analysis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate PARDS
* 3 spontaneous breathing trials failed in less than 7 days

Exclusion Criteria:

* hemodynamic instability
* severe respiratory instability
* contraindication to nasogastric tube exchange
* increase in intracranial pressure
* palliative care for end-stage oncologic disease
* neuromuscular disease
* lesions of medulla

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: during the study, all patients (older than 1 month and younger than 2 years) admitted to Pediatric Intensive Care Unit for moderate pediatric Acute Respiratory Distress Syndrome and ready for weaning from mechanical ventilation were evaluated.
  All patients who failed up to 3 SBTs taking less than 7 days, presenting at least two of the following signs: diaphoresis, nasal flaring, tachycardia (Heart Rate increase ≥ 40 bpm) cardiac arrhythmias, hypotension, apnea, PETCO2 increase > 10 mmHg, decrease of arterial pH < 7.32, PaO2 < 60mmHg with an FiO2 ≥ 0.40 (PaO2/FiO2 less than 150), were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-07-30 (Actual)

PRIMARY OUTCOMES:
asynchrony index | three years
  in each study condition, the asynchrony index was measured. The asynchrnony index value grater than 10% is an indicator of worsening patient-ventilator interaction. the Asynchrony Index is the ratio between the number of asynchronous events and the total respiratory rate, expressed as percentage

SECONDARY OUTCOMES:
patient-ventilator interaction | three years
  the variable describing patient-ventilator interaction is the inspiratory trigger delay (defined as the time lag between the onset of neural inspiration and the onset of ventilatory assistance and measured in milliseconds )
interaction | three years
  another variable describing patient-ventilator interaction is the expiratory trigger delay ( defined as the time lag between the neural expiration and the end of mechanical assistance and measured in milliseconds)
synchrony between patient and mechanical ventilator | three years
  the time of synchrony is the time during which the patient inspiratory effort and the ventilatory assistance are in phase and measured in milliseconds).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio P Conti, Prof, Study Director — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanch L, Villagra A, Sales B, Montanya J, Lucangelo U, Lujan M, Garcia-Esquirol O, Chacon E, Estruga A, Oliva JC, Hernandez-Abadia A, Albaiceta GM, Fernandez-Mondejar E, Fernandez R, Lopez-Aguilar J, Villar J, Murias G, Kacmarek RM. Asynchronies during mechanical ventilation are associated with mortality. Intensive Care Med. 2015 Apr;41(4):633-41. doi: 10.1007/s00134-015-3692-6. Epub 2015 Feb 19. PMID 25693449
- [Background] Blokpoel RG, Burgerhof JG, Markhorst DG, Kneyber MC. Patient-Ventilator Asynchrony During Assisted Ventilation in Children. Pediatr Crit Care Med. 2016 May;17(5):e204-11. doi: 10.1097/PCC.0000000000000669. PMID 26914624
- [Background] Thille AW, Rodriguez P, Cabello B, Lellouche F, Brochard L. Patient-ventilator asynchrony during assisted mechanical ventilation. Intensive Care Med. 2006 Oct;32(10):1515-22. doi: 10.1007/s00134-006-0301-8. Epub 2006 Aug 1. PMID 16896854
- [Background] Bordessoule A, Emeriaud G, Morneau S, Jouvet P, Beck J. Neurally adjusted ventilatory assist improves patient-ventilator interaction in infants as compared with conventional ventilation. Pediatr Res. 2012 Aug;72(2):194-202. doi: 10.1038/pr.2012.64. PMID 22580718
- [Background] Breatnach C, Conlon NP, Stack M, Healy M, O'Hare BP. A prospective crossover comparison of neurally adjusted ventilatory assist and pressure-support ventilation in a pediatric and neonatal intensive care unit population. Pediatr Crit Care Med. 2010 Jan;11(1):7-11. doi: 10.1097/PCC.0b013e3181b0630f. PMID 19593246
- [Background] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Derived] Spinazzola G, Costa R, De Luca D, Chidini G, Ferrone G, Piastra M, Conti G. Pressure Support Ventilation (PSV) versus Neurally Adjusted Ventilatory Assist (NAVA) in difficult to wean pediatric ARDS patients: a physiologic crossover study. BMC Pediatr. 2020 Jul 7;20(1):334. doi: 10.1186/s12887-020-02227-1. PMID 32631305